CLINICAL TRIAL: NCT05403450
Title: A Phase 1-2, Open-Label Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Activity of Tolinapant in Combination With Oral Decitabine/Cedazuridine and Oral Decitabine/Cedazuridine Alone in Subjects With Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: A Study of Tolinapant in Combination With Oral Decitabine/Cedazuridine and Oral Decitabine/Cedazuridine Alone in Participants With Relapsed/Refractory Peripheral T-cell Lymphoma (R/R PTCL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASTX660-03; 2021-005338-40 (EudraCT Number)
Record Dates: First submitted 2022-05-23; First posted 2022-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Relapsed/Refractory Peripheral T-cell Lymphoma
Keywords: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Non-Hodgkin | interventions — ASTX-660; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phases 1 and 2: Tolinapant + Oral Decitabine/Cedazuridine (Experimental): Tolinapant, orally, once daily (QD) on Days 1 to 7 and 15 to 21 of each 28-day cycle in combination with oral decitabine/cedazuridine fixed-dose combination (FDC) tablet, QD on days determined by the Lead-in Phase during each 28-day cycle. The starting dose of tolinapant will be escalated stepwise in successive cohorts until the RP2D is determined.
  Based on RP2D and results determined from Phase 1 participants would receive tolinapant at the identified RP2D in combination with decitabine/cedazuridine, FDC tablet, orally, QD on days determined by the Lead-in Phase during each 28-day cycle in Phase 2.
  Interventions: Drug: Tolinapant; Drug: Decitabine + Cedazuridine
- Phase 1: Oral Decitabine/Cedazuridine (Experimental): Decitabine/cedazuridine FDC tablet, orally, QD on days determined by the Lead-in Phase during each 28-day cycle.
  Interventions: Drug: Decitabine + Cedazuridine

INTERVENTIONS:
Drug: Tolinapant — Capsule for oral administration
  Other Names: ASTX660
  Arms: Phases 1 and 2: Tolinapant + Oral Decitabine/Cedazuridine
Drug: Decitabine + Cedazuridine — Tablet for oral administration
  Other Names: ASTX727

SUMMARY:
The primary purpose of the study is to assess safety, and to identify the recommended phase 2 dose (RP2D) of tolinapant in combination with oral decitabine/cedazuridine in Phase 1 and to assess preliminary efficacy as determined by overall response rate (ORR) in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with expected life expectancy of >12 weeks.
2. Participants must have histologically confirmed R/R PTCL (local pathology report) as defined by 2016 World Health Organization (WHO) classification. The following subtypes are eligible for the study:

   1. Extranodal natural killer (NK)/T-cell lymphoma nasal type.
   2. Enteropathy-associated T-cell lymphoma.
   3. Monomorphic epitheliotropic intestinal T-cell lymphoma.
   4. Hepatosplenic T-cell lymphoma.
   5. Subcutaneous panniculitis-like T-cell lymphoma.
   6. Peripheral T-cell lymphoma not otherwise specified (PTCL-NOS).
   7. Angioimmunoblastic T-cell lymphoma.
   8. Follicular peripheral T-cell lymphoma.
   9. Nodal peripheral T-cell with T-follicular helper (THF) phenotype.
   10. Anaplastic large-cell lymphoma (ALCL).
3. Participants must have evidence of progressive disease and must have received at least two prior systemic therapies.
4. Participants must have measurable disease by contrast-enhanced diagnostic CT (at least 1 nodal lesion >1.5 centimeters (cm) or extranodal lesions >1.0 cm).
5. Participants with CD30-positive disease must have received, be ineligible for, or intolerant to brentuximab vedotin.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Acceptable organ function as per protocol.
8. Women of childbearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.

Exclusion Criteria:

1. Prior treatment with tolinapant or any hypomethylating agent.
2. Hypersensitivity to tolinapant or oral decitabine/cedazuridine, excipients of the drug product, or other components of the study treatment regimen.
3. Poor medical risk because of systemic diseases (e.g., uncontrolled infections) in addition to the qualifying disease under study.
4. Life-threatening illness, significant organ system dysfunction, or other condition that, in the investigator's opinion, could compromise participant safety or the integrity of the study outcomes, or interfere with the absorption or metabolism of tolinapant.
5. A history of, or at risk for, cardiac disease, as evidenced by 1 or more of the following conditions:

   1. Abnormal left ventricular ejection fraction.
   2. Congestive cardiac failure of Grade ≥3.
   3. Unstable cardiac disease.
   4. History or presence of complete left bundle branch block, third-degree heart block, cardiac pacemaker, or clinically significant arrhythmia.
   5. History of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy.
   6. Screening 12-lead electrocardiogram (ECG) with measurable QTc interval of ≥470 milliseconds (msec) (according to either Fridericia's or Bazett's correction).
   7. Any other condition that, in the opinion of the investigator, could put the participant at increased cardiac risk.
6. Known history of human immunodeficiency virus (HIV) infection; or seropositive results consistent with active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
7. Grade 3 or greater neuropathy.
8. Known significant mental illness or other conditions such as active alcohol or other substance abuse that, in the opinion of the investigator, predisposes the participant to high risk of noncompliance with the protocol treatment or assessments.
9. Prior anticancer treatments or therapies within the indicated time window before first dose of study treatment (tolinapant), as follows:

   1. Cytotoxic chemotherapy or radiotherapy within 4 weeks prior.
   2. Monoclonal antibodies within 4 weeks prior.
   3. At least 12 weeks must have elapsed since chimeric antigen receptor T-cell (CAR-T) infusion.
   4. Small molecules or biologics (investigational or approved) within the longer of 3 weeks or 5 half-lives before study treatment.
10. Monoclonal antibody treatment for rheumatologic conditions within 4 weeks of study drug initiation.
11. Concurrent second malignancy currently requiring active therapy, except breast or prostate cancer stable on or responding to endocrine therapy or superficial bladder cancer.
12. Any concurrent second malignancy that is metastatic.
13. Known central nervous system (CNS) lymphoma.
14. Participants with a history of allogeneic transplant are excluded from this study.
15. Autotransplant within 100 days of the first dose of the study drug(s).
16. Systemic corticosteroids >10 mg prednisone equivalent within 7 days of the first dose of study drug(s).
17. Anti-T-cell directed therapy:

    1. Lymphotoxic agents (e.g., anti-CD52) in the past 12 months.
    2. Inhibitory drugs (e.g., calcineurin inhibitors) within 4 weeks of the first dose of study drug(s).
18. Use of a concomitant medication which is a moderate or strong CYP3A4 inhibitor/inducer within 2 weeks of the start of the study.
19. Use of any vaccine within 10 days of the first dose of the study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Dose Limiting Toxicities (DLTs) | Up to 54 months
  This will be evaluated by looking at the number of participants with treatment-related adverse events, serious adverse events (SAEs), and dose-limiting toxicities (DLTs), which are medical problems severe enough to stop study doctors from increasing a treatment dose.
Phase 2: Antitumor Activity Assessed by Overall Response Rate (ORR) Based on 2014 Lugano Classification Using Computerized Tomography (CT) Imaging as the Primary Modality | Up to 54 months

SECONDARY OUTCOMES:
Phase 1: Number of Participants With TEAEs, SAEs and DLTs in the Oral Decitabine/Cedazuridine Arm | Up to 54 months
Ph 1 & 2: AUC: Area Under the Plasma Concentration-Time Curve | Up to 50 months
Ph 1 & 2: Cmax: Maximum Observed Plasma Concentration | Up to 50 months
Ph 1 & 2: Cmin: Minimum Observed Plasma Concentration at Steady State | Up to 50 months
Ph 1 & 2: Tmax: Time to Maximum Observed Plasma Concentration | Up to 50 months
Ph 1 & 2: t½: Apparent Elimination Half-Life | Up to 50 months
Phase 2: Duration of response (DOR) Based on the Lugano Classification Using CT Imaging as the Primary Modality | Up to 54 months
Phase 2: Percentage of Participants With Complete Response (CR) Based on the Lugano Classification Using CT Imaging as the Primary Modality | Up to 54 months
Phase 2: Percentage of Participants With Partial Response (PR) Based on the Lugano Classification Using CT Imaging as the Primary Modality | Up to 54 months
Phase 2: Progression-Free Survival (PFS) Based on the Lugano Classification Using CT Imaging as the Primary Modality | Up to 54 months
Phase 2: Disease Control Rate (DCR) Assessed as Percentage of Participants With Disease Control Based on the Lugano Classification Using CT Imaging as the Primary Modality | Up to 54 months
Phase 2: Overall Survival (OS) Based on the Lugano Classification Using CT Imaging as the Primary Modality | Up to 54 months
Phase 2: Percentage of Participants With DOR, CR, PR, PFS, DCR,and OS Based on the Lugano Classification Using CT Along With PET Imaging Assessments | Up to 54 months
  Duration of response (DOR), complete response (CR), partial response (PR), progression-free survival (PFS), disease control rate (DCR)and overall survival (OS)
Phase 2: Percentage of Participants With Anti-Tumor Activity Based on Assessment Using 2014 Lugano Classification With Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) | Up to 54 months
  Anti-tumor activity in terms of ORR, DOR, CR, PR, and PFS will be evaluated based on assessment using 2014 Lugano Classification with LYRIC.
Phase 2: Percentage of Participants With Anti-Tumor Activity Based on PTCL Subtypes Anti-tumor activity in terms of ORR, DOR, DCR, CR, and PR will be evaluated based on PTCL subtypes (using both pathology and molecular markers). | Up to 54 months

CONTACTS AND LOCATIONS:
Locations (46):
- United States (16):
  - City of Hope Site #151, Duarte, California
  - University of Califonia, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado Anschutz Medical Campus Site #118, Aurora, Colorado
  - Yale Cancer Center Site #109, New Haven, Connecticut
  - Moffitt Cancer Center Site #157, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute Site#159, Detroit, Michigan
  - Rochester Skin Lymphoma Medical Group, PLLC Site #147, Fairport, New York
  - NYU Langone Laura and Isaac Perlmutter Cancer Center Site #153, New York, New York
  - University of Pennsylvania Site# 160, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center Site #101, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (3):
  - Concord Hospital, Concord, New South Wales
  - Monash Medical Center, Melbourne, Victoria
  - Linear Clinical Research Site #834, Nedlands
- France (8):
  - Hôpital Bretonneau, Tours, Indre-et-Loire
  - Centre Henri Becquerel, Rouen, Seine-Maritime
  - Institut Bergonié Site#553, Bordeaux
  - Institut Paoli-Calmettes, Marseille
  - CHU Saint-Eloi Site#556, Montpellier
  - Centre Antoine Lacassagne, Nice
  - AP-HP Pitie Saltpetriere Site# 552, Paris
  - Institut Gustave Roussy, Villejuif
- Italy (6):
  - Ospedale Santa Maria delle Croci di Ravenna, Ravenna, Emilia-Romagna
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forli-Cesena
  - U.O.C. di Ematologia Pad. 8IRCCS Azienda OspedalieroUniversitaria di Bologna Site#651, Bologna
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia Site#650, Brescia
  - Istituto Europeo di Oncologia Site#652, Milan
  - Fondazione IRCCS San Gerardo dei Tintori Site #655, Monza
- Poland (3):
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw, Masovia
  - Ośrodek Badań Klinicznych Wczesnych Faz - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk, Pomeranian Voivodeship
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Lodz, Łódź Voivodeship
- Spain (7):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona, Catalonia
  - Hospital del Mar Site #704, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz Site #703, Madrid
  - Hospital Universitario 12 de Octubre Site#710, Madrid
  - Hospital Universitario Marqués de Valdecilla Site#711, Santander
- United Kingdom (3):
  - Guy's and Saint Thomas' NHS Foundation Trust, London, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England

IPD SHARING:
Plan to Share IPD: No